CLINICAL TRIAL: NCT03584282
Title: Interventions to Improve the HIV PrEP Cascade Among Methamphetamine Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joanne Stekler, MD MPH, Associate Professor, School of Medicine: Allergy and Infectious Diseases, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004760; 1R34DA045620-01 (NIH)
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: HIV/AIDS; Adherence, Medication; Drug Use
Keywords: Pre-Exposure Prophylaxis (PrEP); Methamphetamine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Intervention Model Description: The investigators will randomly assign 10 participants to each arm: 1) standard of care, 2) text messaging only, 3) peer navigation only, and 4) text messaging and peer navigation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (No Intervention): Participants in this group will receive the standard of care for PrEP follow-up and no additional research interventions.
- Text Messaging (Active Comparator): Participants in this group will receive the text messaging intervention.
  Interventions: Behavioral: Text Messaging
- Peer Navigation (Active Comparator): Participants in this group will receive the peer navigator intervention.
  Interventions: Behavioral: Peer Navigation
- Text Messaging and Peer Navigation (Active Comparator): Participants in this group will receive both the text messaging and peer navigation interventions.
  Interventions: Behavioral: Text Messaging; Behavioral: Peer Navigation

INTERVENTIONS:
Behavioral: Text Messaging — The text messaging intervention will send three text messages per day from a library. One will be a reminder to take PrEP, one will include PrEP information, and the third will have the content of the participant's choosing from categories of harm reduction messages and health information. Participants will also select the time period to receive these texts.
  Arms: Text Messaging; Text Messaging and Peer Navigation
Behavioral: Peer Navigation — The peer navigation intervention will provide support from a peer that is responsive to a participant's individualized needs. Peer support may include phone call reminders, help refilling PrEP prescriptions, transit assistance, or other referrals.
  Arms: Peer Navigation; Text Messaging and Peer Navigation

SUMMARY:
Despite increasing knowledge about and use of PrEP nationally, HIV continues to have disproportionate impact among cisgender men and transgender persons who have sex with men and transgender persons (MSM/TG), with methamphetamine (meth)-users being at particularly high risk. Building on their preliminary work, the investigators will pilot text messaging and peer navigation interventions to support PrEP use among meth-using MSM/TG with potential to be cost-effective, scalable, and easily adaptable.

DETAILED DESCRIPTION:
Despite increasing knowledge about and use of PrEP nationally, HIV continues to have disproportionate impact among cisgender men and transgender persons who have sex with men and transgender persons (MSM/TG), with methamphetamine (meth)-users being at particularly high risk. Despite apparent high levels of PrEP knowledge and exceptional insurance and medication coverage, few meth-users in Western WA have enrolled in local PrEP programs. The investigators' preliminary work with meth-using MSM/TG has identified both traditional barriers to PrEP and barriers specific for meth users, including competing priorities (e.g., getting high); lack of regularity in daily schedules leading to difficulties complying with appointments and medication adherence; and concomitant wellness and social concerns, notably depression and meth-related stigma. Additional work is needed to develop new strategies to increase PrEP uptake and support persistence and adherence among meth-using MSM/TG. Building on their preliminary work, the investigators will pilot text messaging and peer navigation interventions to support PrEP use among meth-using MSM/TG with potential to be cost-effective, scalable, and easily adaptable. The first, peer navigation, has been studied in ARV treatment and has been proposed for PrEP. The second, text messaging, has been shown to increase ARV and PrEP adherence.

ELIGIBILITY:
Inclusion Criteria:

* Meets the clinic's eligibility criteria for PrEP
* 18 years of age or older
* HIV-negative
* Cisgender man or individual on the trans gender variant spectrum who has sex with men
* Ability to understand, read, and speak English
* Reports meth use in the past 3 months
* Has a cell phone able to send and receive text messages

Exclusion Criteria:

* PrEP use in the prior month,
* Discomfort or anxiety with regards to text messaging.
* Has any circumstances that, based on the study staff's opinion, would preclude provision of informed consent, make participation unsafe, or make it unlikely the participant would be able to participate for 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender men, transgender women, transgender men, and genderqueer individuals
Enrollment: 21 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Stekler, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Kelley-Ross One-Step PrEP, Seattle, Washington
  - Gay City, Seattle, Washington

REFERENCES:
- [Background] Mera R, McCallister S, Palmer B, Mayer G, Magnuson D, Rawlings K. Truvada (TVD) for HIV pre-exposure prophylaxis (PrEP) utilization in the United States (2013-2015). 21st International AIDS Conference; Durban, South Africa; July 18-22, 2016 [abstract TUAX0105LB]. In.
- [Background] Hood JE, Buskin SE, Dombrowski JC, Kern DA, Barash EA, Katz DA, Golden MR. Dramatic increase in preexposure prophylaxis use among MSM in Washington state. AIDS. 2016 Jan 28;30(3):515-9. doi: 10.1097/QAD.0000000000000937. PMID 26562845
- [Background] Beyrer C, Baral SD, van Griensven F, Goodreau SM, Chariyalertsak S, Wirtz AL, Brookmeyer R. Global epidemiology of HIV infection in men who have sex with men. Lancet. 2012 Jul 28;380(9839):367-77. doi: 10.1016/S0140-6736(12)60821-6. Epub 2012 Jul 20. PMID 22819660
- [Background] Pitasi M, Llata E, Stenger M, Kerani R, Kohn R, Murphy R, et al. HIV prevalence among transgender women and men: results from the STD Surveillance Network, 2010-2013. 2015 National HIV Prevention Conference; Atlanta, GA; December 6-9, 2015 [abstract #1193]. In.
- [Background] Habarta N, Wang G, Mulatu MS, Larish N. HIV Testing by Transgender Status at Centers for Disease Control and Prevention-Funded Sites in the United States, Puerto Rico, and US Virgin Islands, 2009-2011. Am J Public Health. 2015 Sep;105(9):1917-25. doi: 10.2105/AJPH.2015.302659. Epub 2015 Jul 16. PMID 26180964
- [Background] Buskin S, Hood J, Katz DA. Estimating the population-level impact of methamphetamine use on HIV acquisition among men who have sex with men using population attributable risk percent - a powerful and underused planning tool. International AIDS Society Conference 2015. July 19-22, 2015. Vancouver. Abstract MOPEC491. In.
- [Background] McMahan V, Martin A, Garske L, Baeten JM, Banta-Green C, Stekler J. Knowledge about PrEP among MSM and Trans* Methamphetamine Users in Seattle. 24th Conference on Retroviruses and Opportunistic Infections; Seattle, WA; February 13-16, 2017 [#2063]. In.
- [Background] Simoni JM, Huh D, Frick PA, Pearson CR, Andrasik MP, Dunbar PJ, Hooton TM. Peer support and pager messaging to promote antiretroviral modifying therapy in Seattle: a randomized controlled trial. J Acquir Immune Defic Syndr. 2009 Dec 1;52(4):465-473. doi: 10.1097/qai.0b013e3181b9300c. PMID 19911481
- [Background] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Background] Dowshen N, Kuhns LM, Johnson A, Holoyda BJ, Garofalo R. Improving adherence to antiretroviral therapy for youth living with HIV/AIDS: a pilot study using personalized, interactive, daily text message reminders. J Med Internet Res. 2012 Apr 5;14(2):e51. doi: 10.2196/jmir.2015. PMID 22481246
- [Background] Finitsis DJ, Pellowski JA, Johnson BT. Text message intervention designs to promote adherence to antiretroviral therapy (ART): a meta-analysis of randomized controlled trials. PLoS One. 2014 Feb 5;9(2):e88166. doi: 10.1371/journal.pone.0088166. eCollection 2014. PMID 24505411
- [Background] Liu A, Stojanovski K, Lester R. Developing and Implementing a Mobile Health (mHealth) Adherence Support System for HIV- Uninfected Men who have Sex with Men (MSM) Taking Pre-Exposure Prophylaxis (PrEP): The iText Study. 8th International Conference on HIV Treatment and Prevention Adherence; Miami, FL; June 2-4, 2013 [Abstract #165]. In.
- [Derived] Frank N, McMahan VM, Violette LR, Martin A, Glick SN, Stekler JD. Efficient Expansion of a Behavioral Survey to Assess Sex, Gender, and Behavioral Risk Among Transgender and Nonbinary Individuals: HMU! (HIV Prevention for Methamphetamine Users). Transgend Health. 2023 Oct 4;8(5):472-476. doi: 10.1089/trgh.2021.0082. eCollection 2023 Oct. PMID 37810934
- [Derived] McMahan VM, Frank N, Buckler S, Violette LR, Baeten JM, Banta-Green CJ, Barnabas RV, Simoni J, Stekler JD. Protocol Development for HMU! (HIV Prevention for Methamphetamine Users), a Study of Peer Navigation and Text Messaging to Promote Pre-Exposure Prophylaxis Adherence and Persistence Among People Who Use Methamphetamine: Qualitative Focus Group and Interview Study. JMIR Form Res. 2020 Sep 14;4(9):e18118. doi: 10.2196/18118. PMID 32924952

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care/Text Messaging: Participants in this group will receive the standard of care the text messaging intervention.
  Text Messaging: The text messaging intervention will send three text messages per day from a library. One will be a reminder to take PrEP, one will include PrEP information, and the third will have the content of the participant's choosing from categories of harm reduction messages and health information. Participants will also select the time period to receive these texts.
  Study intervention groups changed over time - the original study design was a 2 x 2 factorial design with peer navigation, text messaging, both interventions, and standard of care arms. However, with slow enrollment, reports of text messaging being a possible barrier to enrollment, and a smaller anticipated effect compared to peer navigation, the intervention groups were collapsed to a comparison of peer navigation (whether or not text messaging was included) compared to standard of care.
Period: Overall Study
Arm/Group | Standard of Care/Text Messaging | Peer Navigation
Started | 12 | 9
Completed | 5 | 6
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care/Text Messaging | Peer Navigation | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [28 to 40] | 33 [29 to 40] | 35 [29 to 40]
Sex/Gender, Customized [Number; unit: participants]
  cisgender man | 10 | 8 | 18
  transgender female | 1 | 1 | 2
  Non-binary/genderqueer | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  Multiracial | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Text Messaging
Description: Self-reported likelihood to recommend the text messaging intervention, via survey response, among those who received the text messaging intervention (may have been in the Standard of care group or the Peer Navigation group). Only participants who received the text messaging intervention are included in the analysis group.
Time Frame: 6 months
Population: Self-reported likelihood to recommend the text messaging intervention, via survey response, among those who received the text messaging intervention (may have been in the Standard of care group or the Peer Navigation group). Only participants who received the text messaging intervention are included in the analysis group.
Measure: Count of Participants; unit: Participants
Groups:
- Peer Navigation: Participants in this group will receive the peer navigator intervention. Some were also assigned text messaging.
  Peer Navigation: The peer navigation intervention will provide support from a peer that is responsive to a participant's individualized needs. Peer support may include phone call reminders, help refilling PrEP prescriptions, transit assistance, or other referrals.
Arm/Group | Standard of Care/Text Messaging | Peer Navigation
Number analyzed (Participants) | 3 | 3
Participants
  Very Unlikely to Recommend | 0 | 0
  Unlikely to Recommend | 0 | 1
  Neither Unlikely nor Likely to Recommend | 1 | 0
  Likely to Recommend | 0 | 0
  Very Likely to Recommend | 1 | 1
  Data Missing (e.g. Survey not completed, question left blank) | 1 | 1

2. Secondary Outcome: PrEP Persistence
Description: Persistence on PrEP comparing standard of care or text messaging vs peer navigation, as measured by whether the participant had returned to the clinic at 6 months follow up their DBS card collection.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care/Text Messaging | Peer Navigation
Number analyzed (Participants) | 12 | 9
Participants | 4 | 6

3. Secondary Outcome: PrEP Adherence
Description: PrEP adherence measured in dried blood spots comparing standard of care/text messaging vs peer navigation, as measured by the detection of tenofovir-diphosphate (TFV-DP) in DBS collected 6 months after study enrollment.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care/Text Messaging | Peer Navigation
Number analyzed (Participants) | 12 | 9
Participants
  BLQ | 0 | 1
  <2 doses/week | 1 | 1
  2-3 doses/week | 1 | 1
  4-6 doses/week | 0 | 2
  7 doses/week | 2 | 1
  No DBS collected | 8 | 3

4. Primary Outcome: Acceptability of Peer Navigation
Description: Self-reported likelihood to recommend the peer navigation intervention, via survey response, among those who were assigned to the peer navigation group. Only participants who received the peer navigation intervention are included in the analysis group.
Time Frame: 6 months
Population: Self-reported likelihood to recommend the peer navigation intervention, via survey response, among those who were assigned to the peer navigation group. Only participants who received the peer navigation intervention are included in the analysis group.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Navigation
Number analyzed (Participants) | 9
Participants
  Very Unlikely to Recommend | 0
  Unlikely to Recommend | 0
  Neither Unlikely nor Likely to Recommend | 0
  Likely to Recommend | 1
  Very Likely to Recommend | 3
  Data Missing (e.g. Survey not completed or question left blank) | 5

ADVERSE EVENTS:
Time Frame: 6 months of follow up for each participant, or until loss to follow up.
Arm/Group | Standard of Care/Text Messaging | Peer Navigation
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

LIMITATIONS AND CAVEATS:
Data collected via surveys may have been impacted by social desirability bias. While the HMU! cohort represented some populations disproportionately impacted by methamphetamine and HIV, there were key populations we did not reach. Alaskan Native and Native American and Hispanic/Latinx MSM were under represented in our study, as were individuals who were not cisgender.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03584282/Prot_000.pdf
  • Informed Consent Form (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT03584282/ICF_001.pdf